CLINICAL TRIAL: NCT04977115
Title: Comparison of Intraocular Caliper-assisted and Verion Navigation System-assisted Capsulotomy in Phacoemulsification Surgery: A Randomized Non-inferiority Trial
Brief Title: Clinical Evaluation of Intraocular Caliper-assisted Capsulotomy for Age-related Cataract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021KYPJ110
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraocular caliper-assisted capsulotomy group (Experimental): In intraocular caliper-assisted capsulotomy group, a modified intraocular caliper with standard calibration on the rinse needle was used to measure and locate the position of capsulorhexis with 5.3 mm diameter and the principle of pupillary margin in concentric circles. The surgeon could gently use the blunt needle in the front of the intraocular caliper to further make corresponding markers on the lens anterior capsule, and then carry out capsulotomy according to the marks.
  Interventions: Procedure: Intraocular caliper-assisted capsulotomy
- Verion navigation system-assisted capsulotomy group (Active Comparator): In the Verion-assisted capsulotomy group, Verion navigation system was applied to project a 5.3 mm capsulorhexis centered on the corneal vertex. According to the projected capsulorhexis, capsulotomy was performed.
  Interventions: Procedure: Verion navigation system-assisted capsulotomy

INTERVENTIONS:
Procedure: Intraocular caliper-assisted capsulotomy — Intraocular caliper is a modified intraocular caliper with standard calibration on the rinse needle.
  Arms: Intraocular caliper-assisted capsulotomy group
Procedure: Verion navigation system-assisted capsulotomy — Verion Image Guided System (Alcon Laboratories, Inc.) is a digital image guidance system consisting of a diagnostic reference unit and a surgery pilot for intraoperative surgical assistance. The device can be used to align toric intraocular lens during surgery as well as support manual creation of a capsulorhexis with a predefined target diameter.
  Arms: Verion navigation system-assisted capsulotomy group

SUMMARY:
The purpose of this study is to compare the accuracy of capsulotomy assisted by intraocular caliper and Verion navigation system in phacoemulsification surgery and postoperative visual quality of patients.

DETAILED DESCRIPTION:
Continuous curvilinear capsulorhexis (CCC) is an important and technically challenging procedure in cataract surgery. However, most surgeons perform CCC by experience or referring to the pupil size, which is highly subjective and the accuracy of capsulorhexis is unsatisfactory. The investigators developed a new modified intraocular caliper with standard calibration on the rinse needle, which can measure and locate the position of capsulorhexis. The surgeon can gently use the blunt needle in the front of the intraocular caliper to further make corresponding markers on the lens anterior capsule, and then carry out capsulotomy according to the marks. We found intraocular caliper-assisted capsulotomy can obviously improve the accuracy of capsulorhexis. The purpose of this study is to compare the accuracy and postoperative visual quality of intraocular caliper-assisted capsulotomy with those of digital image projection device VERION navigation system.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 55 to 80 years with age-related cataract;
* Pupil diameter ≥ 6.5mm after pupil dilation;
* Lens nuclear opacity grading score (LOCS III) lower than 4.0.

Exclusion Criteria:

* Patients had previous intraocular surgery;
* Patients with a diagnosed eye disease that may affect the functions of lens suspensory ligament such as previous ocular trauma, lens subluxation, pseudoexfoliation syndrome, retinal pigment degeneration;
* Patients had other ocular diseases that impair visual function include optic neuropathy, uveitis, and tumor.
* Refused to participate the study.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2021-07-26 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Deviation of horizontal and vertical diameter of capsulorhexis from the target diameter (5.3 mm) | During the surgery
  Images of the edges of IOL and capsulorhexis are taken at the end of the operation. Image J image analysis software is used to measure the horizontal diameter and vertical diameter of capsulorhexis with the diameter of IOL optical surface (6 mm) as the reference by two independently professional graders at the meantime, and further calculate the deviation of horizontal and vertical diameter of capsulorhexis from the target diameter (5.3 mm) .

SECONDARY OUTCOMES:
Uncorrected and corrected visual acuity | One month after surgery
  Visual acuity is evaluated with ETDRS visual acuity chart.
Ideal ratio of capsulorhexis | During the surgery
  Ideal capsulorhexis is defined as a centered and round capsulorhexis, which can cover the edge of IOL optical surface continuously for 360 degrees with a diameter between 5.0 to 5.5 mm.
Grades of capsulorhexis-IOL overlap | During the surgery
  The capsulorhexis-IOL overlap of each patient is graded as 360-degree continuous overlap, 270~360-degree overlap, 180~270-degree overlap, 90~180-degree overlap, and < 90-degree overlap.
Distance between pupil center and capsulorhexis center | During the surgery
  Measured by Image J image analysis software.
Horizontal and vertical diameter of capsulorhexis | During the surgery
  Measured by Image J image analysis software.
Intraocular lens tilt | One month after surgery
  Measured by anterior segment OCT (CASIA2).
Intraocular lens decentration | One month after surgery
  Measured by anterior segment OCT (CASIA2).
Intraocular aberrations | One month after surgery
  Measured by OPD-SCAN III.
Deviation of horizontal and vertical diameter of capsulorhexis from the target diameter (5.3 mm) | One month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center，Sun Yat-Sen University, Guangzhou, China

REFERENCES:
- [Derived] Chen X, Liu Z, Jin L, Zheng Y, Luo L, Liu Y. Manual Marking Guidance vs Digital Guidance System-Assisted Capsulorhexis in Phacoemulsification: A Noninferiority Randomized Clinical Trial. JAMA Ophthalmol. 2025 Nov 13. doi: 10.1001/jamaophthalmol.2025.4448. Online ahead of print. PMID 41231447